CLINICAL TRIAL: NCT01522235
Title: A Double-blind, Randomized, Placebo-controlled Trial to Evaluate the Efficacy of Intravenous Immunoglobulin Therapy in Autoimmune Autonomic Ganglionopathy.
Brief Title: Evaluating the Effectiveness of Intravenous Immunoglobulin Therapy in Autoimmune Autonomic Ganglionopathy
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Collaborators: Mayo Clinic (Other); Vanderbilt University (Other); NYU Langone Health (Other); University of Texas Southwestern Medical Center (Other); National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Principal Investigator, Roy Freeman, MD, Professor of Neurology, Harvard Medical School, Beth Israel Deaconess Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2011P000397; 1U54NS065736 (NIH)
Record Dates: First submitted 2012-01-25; First posted 2012-01-31 (Estimated); Results first posted 2017-07-02 (Actual); Last update posted 2017-07-02 (Actual); Status verified 2017-06

CONDITIONS: Autoimmune Autonomic Ganglionopathy (AAG)
Keywords: Autoimmune autonomic neuropathy; Orthostatic hypotension; Dysautonomia; Autonomic failure; Peripheral autonomic neuropathy
MeSH Terms: conditions — Hypotension, Orthostatic; Autonomic Nervous System Diseases; Pure Autonomic Failure | interventions — Immunoglobulins, Intravenous

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: To prevent unblinding because of observed efficacy, adverse events or changes in laboratory values, each site will have both a treating investigator and an examining investigator. The treating investigator will assess the participant's clinical response and laboratory findings. The treating investigator will make all clinical treatment decisions. The examining investigator will monitor only the clinical autonomic symptoms and quality of life scores, and autonomic tests. Both the treating and examining investigators should be physicians. To prevent infusion unblinding, infusions of IVIG and placebo will occur in opaque bags.
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- IVIg group (Active Comparator): Double blinded IVIg and single blinded IVIg
  Interventions: Drug: Double blinded IVIg; Other: Single Blinded IVIg
- Placebo Group (Other): Double blinded Placebo and single blinded IVIg
  Interventions: Other: Double blinded Placebo; Other: Single Blinded IVIg

INTERVENTIONS:
Drug: Double blinded IVIg — Participants will receive study treatment with IVIg, at 2.0 gm/kg over 2-4 consecutive days. A maintenance study treatment IVIg, at 1.0 gm/kg, over 1-2 consecutive days will occur three weeks later. All participants will proceed to the single blind Second Observation Period.
  Other Names: Gammagard
  Arms: IVIg group
Other: Double blinded Placebo — Participants will receive placebo (5% albumin) at 2.0 gm/kg over 2-4 consecutive days. A maintenance treatment with placebo (5% albumin) at 1.0 gm/kg, over 1-2 consecutive days will occur three weeks later. All participants will proceed to the single blind Second Observation Period.
  Arms: Placebo Group
Other: Single Blinded IVIg — This is the single blind Second Observation Period. All participants will receive study treatment with IVIg, at 2.0 gm/kg over 2-4 consecutive days. A maintenance study treatment at 1.0 gm/kg, over 1-2 consecutive days will occur three weeks later.

SUMMARY:
The purpose of the study is to see if administering intravenous immune globulin (IVIG) (putting immune globulin directly into your blood) helps to improve the symptoms of orthostatic hypotension (sudden fall in blood pressure when a person stands up) and quality of life in men and women who have autoimmune autonomic ganglionopathy (AAG).

DETAILED DESCRIPTION:
Autoimmune autonomic ganglionopathy (AAG) is a rare disease that results in severe dysautonomia (disorder of autonomic nervous system function). Many patients are unable to carry out activities of daily living due to autonomic symptoms that do not respond well to therapy (such as drops in blood pressure while standing). The recent discovery of antibodies that cause AAG has stimulated interest in immunomodulatory therapy (therapies that modify the functioning of the immune system). Studies in which a positive clinical response to these therapies have been reported in patients with AAG using immunomodulatory therapy as a treatment.

The investigators plan to carry out a blinded, randomized trial using IVIG. There have been no reported randomized clinical trials with any immunosuppressive agent in AAG. The proposed studies, if successful, will provide the first reliable clinical evidence, that therapy with IVIG is an effective treatment of AAG.

Treatment for the symptoms of autonomic failure is only effective in mild cases. Most patients require therapy that would change the course of the disease, but at present there is no established therapeutic regimen. The natural course of untreated AAG is not known.

To address these unresolved issues, this clinical trial has the following goals:

1. To measure the effect of IVIG treatment on orthostatic hypotension, autonomic symptoms and quality of life scores in patient participants with AAG.
2. To determine the durability of IVIG (how long the treatment is effective) on orthostatic hypotension, autonomic symptoms and quality of life scores in patient participants with AAG.

Participants enrolled in the study will receive two courses of intravenous immunoglobulin or placebo separated by 3 weeks. During the First Observation Period, participants will be evaluated after 6 weeks to determine the clinical response and natural history of the disorder.

All the participants will then move to a single blinded second observation period.

All patients enrolled in the study (IVIG group and placebo group) will receive two infusions of intravenous immunoglobulin, i.e., both cohorts will receive IVIG (although participants will not know this, and physicians will not be aware if this treatment is to IVIG naïve or IVIG continued participants).

ELIGIBILITY:
Inclusion Criteria:

1. Participants aged 18 to 85
2. Participants have neurogenic orthostatic hypotension (fall in systolic blood pressure > 30 mmHg).
3. Symptoms of orthostatic intolerance.
4. Antibodies to the neuronal AChR of the autonomic ganglia of >0.2nmol/l. Results must be within 6 months of the screening visit and there may not have been any immunomodulatory interventions since the time of the antibody measurement or the sample will need to be reconfirmed at screening.
5. Participants must be willing to withdraw from medications that affect vasoactive and autonomic function for 5 half-lives during testing (with the exception of stable doses of fludrocortisone up to 0.2 mg/day) and adhere to a regular diet

Exclusion Criteria:

1. Women of childbearing potential (WOCP) who are not using a medically accepted contraception
2. Pregnant or lactating females- if participants become pregnant during the trial they will no longer receive IVIG, but will be followed as part of the intention to treat protocol.
3. Severe depression and/or anxiety (score of > 29 on the Beck Depression Inventory or score on the Beck Anxiety Inventory of ≥ 36)
4. Active psychosis is ineligible, history of psychosis will be eligible, but only after review with the patients PCP and/or treating mental health provider.
5. History of asthma
6. Other causes of autonomic failure (e.g., diabetes, amyloidosis)
7. History of allergic or anaphylactic reaction to humanized or murine antibodies.
8. History or presence of recurrent or chronic infection (recurrent infections defined as >4 times per year).
9. History of cancer, including solid tumors and hematologic malignancies (except fully resolved and resected cutaneous basal cell and squamous cell carcinomas of the skin)
10. History or presence of vascular disease potentially affecting brain or spinal cord (e.g., stroke, transient ischemic attack, carotid stenosis (greater than 80%), aortic aneurysm, intracranial aneurysm, hemorrhage, arteriovenous malformation)
11. History of severe, clinically significant central nervous system trauma (e.g., cerebral contusion, spinal cord compression)
12. History or presence of infectious causes of encephalopathy or myelopathy (e.g., syphilis, Lyme disease, human T-cell lymphotropic virus type 1 [HTLV-1], herpes zoster myelopathy)
13. History of thromboembolic events or deep vein thrombosis
14. Platelet count <100,000/mL, Hemoglobin <8.5 g/dL, Neutrophils <1.5 x 103/mL.
15. Serum IgA deficiency: Immunoglobulin A (IgA) level < 7 mg/dL.
16. History of immunosuppression or HIV/AIDS
17. History of cardiac arrhythmia or angina, electrocardiogram (ECG) showing significant abnormality that the treating investigator determines may jeopardize the participant's health (i.e., acute ischemia, left bundle branch, or bifascicular block)
18. History of renal failure or creatinine >2.0
19. History of previous allergic response to albumin.
20. Treatment with IVIG or plasma exchange within 6 weeks of study enrollment.
21. Active adjustments of other immunomodulatory treatments. Patients that are on stable doses of immunomodulatory medications (no dose changes within 4 months -including, but not limited to prednisone, mycophenolate mofetil or azathioprine) but still have elevated antibody titers and meet criteria for inclusion will be allowed to participate in the study.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2012-02; Primary Completion 2014-05 (Actual); Study Completion 2015-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Roy Freeman, MD, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (6):
- United States (6):
  - Nih Ninds, Bethesda, Maryland
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - NYU Medical Center, New York, New York
  - Vanderbilt University, Nashville, Tennessee
  - UT Southwestern Medical Center, Dallas, Texas

IPD SHARING:
Plan to Share IPD: Yes
The investigators will adhere to the NIH Grant Policy on Sharing of Unique Research Resources including the Principles and Guidelines for Recipients of NIH Research Grants and Contracts on Obtaining and Disseminating Biomedical Research Resources.

REFERENCES:
- [Background] Vernino S, Sandroni P, Singer W, Low PA. Invited Article: Autonomic ganglia: target and novel therapeutic tool. Neurology. 2008 May 13;70(20):1926-32. doi: 10.1212/01.wnl.0000312280.44805.5d. PMID 18474849
- [Background] Vernino S, Low PA, Fealey RD, Stewart JD, Farrugia G, Lennon VA. Autoantibodies to ganglionic acetylcholine receptors in autoimmune autonomic neuropathies. N Engl J Med. 2000 Sep 21;343(12):847-55. doi: 10.1056/NEJM200009213431204. PMID 10995864
- [Background] Gibbons CH, Freeman R. Antibody titers predict clinical features of autoimmune autonomic ganglionopathy. Auton Neurosci. 2009 Mar 12;146(1-2):8-12. doi: 10.1016/j.autneu.2008.11.013. Epub 2009 Jan 13. PMID 19144572
- [Background] Klein CM, Vernino S, Lennon VA, Sandroni P, Fealey RD, Benrud-Larson L, Sletten D, Low PA. The spectrum of autoimmune autonomic neuropathies. Ann Neurol. 2003 Jun;53(6):752-8. doi: 10.1002/ana.10556. PMID 12783421
- [Background] Gibbons CH, Vernino SA, Kaufmann H, Freeman R. L-DOPS therapy for refractory orthostatic hypotension in autoimmune autonomic neuropathy. Neurology. 2005 Oct 11;65(7):1104-6. doi: 10.1212/01.wnl.0000178980.83477.14. PMID 16217067
- [Background] Gibbons CH, Vernino SA, Freeman R. Combined immunomodulatory therapy in autoimmune autonomic ganglionopathy. Arch Neurol. 2008 Feb;65(2):213-7. doi: 10.1001/archneurol.2007.60. PMID 18268189
- [Background] Iodice V, Kimpinski K, Vernino S, Sandroni P, Fealey RD, Low PA. Efficacy of immunotherapy in seropositive and seronegative putative autoimmune autonomic ganglionopathy. Neurology. 2009 Jun 9;72(23):2002-8. doi: 10.1212/WNL.0b013e3181a92b52. PMID 19506222
- [Background] Modoni A, Mirabella M, Madia F, Sanna T, Lanza G, Tonali PA, Silvestri G. Chronic autoimmune autonomic neuropathy responsive to immunosuppressive therapy. Neurology. 2007 Jan 9;68(2):161-2. doi: 10.1212/01.wnl.0000251194.82212.75. No abstract available. PMID 17210903
- [Background] Young RR, Asbury AK, Adams RD, Corbett JL. Pure pan-dysautonomia with recovery. Trans Am Neurol Assoc. 1969;94:355-7. No abstract available. PMID 5374487
- [Background] Vernino S, Ermilov LG, Sha L, Szurszewski JH, Low PA, Lennon VA. Passive transfer of autoimmune autonomic neuropathy to mice. J Neurosci. 2004 Aug 11;24(32):7037-42. doi: 10.1523/JNEUROSCI.1485-04.2004. PMID 15306637
- [Background] Malik U, Oleksowicz L, Latov N, Cardo LJ. Intravenous gamma-globulin inhibits binding of anti-GM1 to its target antigen. Ann Neurol. 1996 Jan;39(1):136-9. doi: 10.1002/ana.410390121. PMID 8572660
- [Background] Kazatchkine MD, Kaveri SV. Immunomodulation of autoimmune and inflammatory diseases with intravenous immune globulin. N Engl J Med. 2001 Sep 6;345(10):747-55. doi: 10.1056/NEJMra993360. No abstract available. PMID 11547745
- [Background] Dalakas MC. Intravenous immunoglobulin in autoimmune neuromuscular diseases. JAMA. 2004 May 19;291(19):2367-75. doi: 10.1001/jama.291.19.2367. PMID 15150209
- [Background] Samuelsson A, Towers TL, Ravetch JV. Anti-inflammatory activity of IVIG mediated through the inhibitory Fc receptor. Science. 2001 Jan 19;291(5503):484-6. doi: 10.1126/science.291.5503.484. PMID 11161202
- [Background] Dalakas MC. Blockade of blocking antibodies in Guillain-Barre syndromes: "unblocking" the mystery of action of intravenous immunoglobulin. Ann Neurol. 2002 Jun;51(6):667-9. doi: 10.1002/ana.10259. No abstract available. PMID 12112069
- [Background] Hughes RA, Cornblath DR. Guillain-Barre syndrome. Lancet. 2005 Nov 5;366(9497):1653-66. doi: 10.1016/S0140-6736(05)67665-9. PMID 16271648
- [Background] Eftimov F, Winer JB, Vermeulen M, de Haan R, van Schaik IN. Intravenous immunoglobulin for chronic inflammatory demyelinating polyradiculoneuropathy. Cochrane Database Syst Rev. 2013 Dec 30;(12):CD001797. doi: 10.1002/14651858.CD001797.pub3. PMID 24379104
- [Background] Leger JM, Viala K, Cancalon F, Maisonobe T, Gruwez B, Waegemans T, Bouche P. Intravenous immunoglobulin as short- and long-term therapy of multifocal motor neuropathy: a retrospective study of response to IVIg and of its predictive criteria in 40 patients. J Neurol Neurosurg Psychiatry. 2008 Jan;79(1):93-6. doi: 10.1136/jnnp.2007.121756. PMID 18079302
- [Background] Slee M, Selvan A, Donaghy M. Multifocal motor neuropathy: the diagnostic spectrum and response to treatment. Neurology. 2007 Oct 23;69(17):1680-7. doi: 10.1212/01.wnl.0000277697.55288.d0. PMID 17954783
- [Background] Federico P, Zochodne DW, Hahn AF, Brown WF, Feasby TE. Multifocal motor neuropathy improved by IVIg: randomized, double-blind, placebo-controlled study. Neurology. 2000 Nov 14;55(9):1256-62. doi: 10.1212/wnl.55.9.1256. PMID 11087764
- [Background] Gorson KC, Ropper AH, Weinberg DH, Weinstein R. Efficacy of intravenous immunoglobulin in patients with IgG monoclonal gammopathy and polyneuropathy. Arch Neurol. 2002 May;59(5):766-72. doi: 10.1001/archneur.59.5.766. PMID 12020258
- [Background] Zinman L, Ng E, Bril V. IV immunoglobulin in patients with myasthenia gravis: a randomized controlled trial. Neurology. 2007 Mar 13;68(11):837-41. doi: 10.1212/01.wnl.0000256698.69121.45. PMID 17353471
- [Background] Maddison P, Newsom-Davis J. Treatment for Lambert-Eaton myasthenic syndrome. Cochrane Database Syst Rev. 2005 Apr 18;(2):CD003279. doi: 10.1002/14651858.CD003279.pub2. PMID 15846654
- [Background] Dalakas MC, Illa I, Dambrosia JM, Soueidan SA, Stein DP, Otero C, Dinsmore ST, McCrosky S. A controlled trial of high-dose intravenous immune globulin infusions as treatment for dermatomyositis. N Engl J Med. 1993 Dec 30;329(27):1993-2000. doi: 10.1056/NEJM199312303292704. PMID 8247075
- [Background] Gold R, Dalakas MC, Toyka KV. Immunotherapy in autoimmune neuromuscular disorders. Lancet Neurol. 2003 Jan;2(1):22-32. doi: 10.1016/s1474-4422(03)00264-3. PMID 12849298
- [Background] Linker RA, Gold R. Use of intravenous immunoglobulin and plasma exchange in neurological disease. Curr Opin Neurol. 2008 Jun;21(3):358-65. doi: 10.1097/WCO.0b013e3282ff5b8f. PMID 18451723
- [Background] Donofrio PD, Berger A, Brannagan TH 3rd, Bromberg MB, Howard JF, Latov N, Quick A, Tandan R. Consensus statement: the use of intravenous immunoglobulin in the treatment of neuromuscular conditions report of the AANEM ad hoc committee. Muscle Nerve. 2009 Nov;40(5):890-900. doi: 10.1002/mus.21433. PMID 19768755
- [Background] Heafield MT, Gammage MD, Nightingale S, Williams AC. Idiopathic dysautonomia treated with intravenous gammaglobulin. Lancet. 1996 Jan 6;347(8993):28-9. doi: 10.1016/s0140-6736(96)91559-7. PMID 8531546
- [Background] Mericle RA, Triggs WJ. Treatment of acute pandysautonomia with intravenous immunoglobulin. J Neurol Neurosurg Psychiatry. 1997 May;62(5):529-31. doi: 10.1136/jnnp.62.5.529. PMID 9153616

RESULTS

PARTICIPANT FLOW:
Groups:
- IVIG Group: IVIg
  IVIg: Participants will receive study treatment with IVIg, at 2.0 gm/kg over 2-4 consecutive days. A maintenance study treatment IVIg, at 1.0 gm/kg, over 1-2 consecutive days will occur three weeks later. All participants will proceed to the single blind Second Observation Period.
- Placebo Group: Placebo
  2 treatments of placebo and 2 treatments of IVIg: Participants will receive placebo (5% albumin) at 2.0 gm/kg over 2-4 consecutive days. A maintenance treatment with placebo (5% albumin) at 1.0 gm/kg, over 1-2 consecutive days will occur three weeks later. All participants will proceed to the single blind Second Observation Period.
Period: Overall Study
Arm/Group | IVIG Group | Placebo Group
Started | 3 | 3
Randomized | 2 | 3
Completed | 2 | 2
Not Completed | 1 | 1
Not completed — Physician Decision | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Group A: IVIg
  IVIG: Participants will receive study treatment with IVIg, at 2.0 gm/kg over 2-4 consecutive days. A maintenance study treatment IVIg, at 1.0 gm/kg, over 1-2 consecutive days will occur three weeks later. All participants will proceed to the single blind Second Observation Period.
  They will receive study treatment with IVIg, at 2.0 gm/kg over 2-4 consecutive days. A maintenance study treatment at 1.0 gm/kg, over 1-2 consecutive days will occur three weeks later.
- Group B: Placebo
  2 treatments of placebo and 2 treatments of IVIg: Participants will receive placebo (5% albumin) at 2.0 gm/kg over 2-4 consecutive days. A maintenance treatment with placebo (5% albumin) at 1.0 gm/kg, over 1-2 consecutive days will occur three weeks later. All participants will proceed to the single blind Second Observation Period.
  They will receive study treatment with IVIg, at 2.0 gm/kg over 2-4 consecutive days. A maintenance study treatment at 1.0 gm/kg, over 1-2 consecutive days will occur three weeks later.
- Total: Total of all reporting groups
Arm/Group | Group A | Group B | Total
Number analyzed (Participants) | 3 | 3 | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 3 | 3 | 6
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 3 | 4
  Male | 2 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Change in Systolic Blood Pressure During 60° Tilt (ΔSBP)
Description: The primary outcome, the change in systolic blood pressure during 60 degree tilt (ΔSBP), will be assessed in all study participants at baseline and at 6 weeks.
Time Frame: Baseline and 6 weeks
Measure: Mean (Standard Deviation); unit: mmHg
Groups:
- IVIg Group: IVIg
  IVIg: Participants will receive study treatment with IVIg, at 2.0 gm/kg over 2-4 consecutive days. A maintenance study treatment IVIg, at 1.0 gm/kg, over 1-2 consecutive days will occur three weeks later. All participants will proceed to the single blind Second Observation Period.
  They will receive study treatment with IVIg, at 2.0 gm/kg over 2-4 consecutive days. A maintenance study treatment at 1.0 gm/kg, over 1-2 consecutive days will occur three weeks later.
- Placebo Group: Placebo
  2 treatments of placebo and 2 treatments of IVIG: Participants will receive placebo (5% albumin) at 2.0 gm/kg over 2-4 consecutive days. A maintenance treatment with placebo (5% albumin) at 1.0 gm/kg, over 1-2 consecutive days will occur three weeks later. All participants will proceed to the single blind Second Observation Period.
  They will receive study treatment with IVIg, at 2.0 gm/kg over 2-4 consecutive days. A maintenance study treatment at 1.0 gm/kg, over 1-2 consecutive days will occur three weeks later.
Arm/Group | IVIg Group | Placebo Group
Number analyzed (Participants) | 2 | 3
mmHg | 42.5 (54.4) | -12.3 (38.0)

2. Secondary Outcome: Change in Systolic Blood Pressure During 60° Tilt (ΔSBP)
Description: To compare the change in systolic blood pressure during 60 degree head up tilt table test after 6 and 12 weeks of IVIG (the within-patient difference in ΔSBP at 12 and 6 weeks among treated patients).
Time Frame: 6 weeks and 12 weeks
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | IVIG Group | Placebo Group
Number analyzed (Participants) | 2 | 3
mmHg | -26 (43.8) | -7.6 (7.09)

3. Secondary Outcome: Composite Autonomic Symptom Score [COMPASS] Questionnaire
Description: To determine the change in autonomic symptoms (measured by the composite autonomic symptom score [COMPASS] questionnaire) measured at baseline and 6 weeks. Minimum and maximum score possible: 0-100. We have reported the Total score. Higher values represent worse outcome.
Time Frame: Baseline, 6 weeks
Measure: Mean (Standard Deviation); unit: units
Arm/Group | IVIg Group | Placebo Group
Number analyzed (Participants) | 2 | 3
units | -5 (2.8) | -0.33 (5.13)

4. Secondary Outcome: Composite Autonomic Severity Score (CASS) Questionnaire.
Description: To determine the change in autonomic symptoms (measured by the composite autonomic severity score [CASS]) measured at baseline and 6 weeks in individuals receiving IVIg.
  Is a 10-point composite autonomic scoring scale of autonomic function. This scale allots 4 points for adrenergic and 3 points each for sudomotor and cardiovagal failure. Subjects with a score of 3 or less on have a mild autonomic failure, 4-6 have moderate autonomic failure and those with scores of 7 to 10 have severe failure. The minimum score possible is 3 and maximum is 10.
Time Frame: Baseline, 6 weeks
Measure: Mean (Standard Deviation); unit: units
Arm/Group | IVIg Group | Placebo Group
Number analyzed (Participants) | 2 | 3
units | 0.5 (0.7) | 0 (0)

5. Secondary Outcome: EuroQol [EQ-5D] Questionnaire.
Description: To determine the change in quality of life (measured by the EuroQol [EQ-5D]) measured at baseline and 6 weeks in individuals receiving IVIg. We have reported the subscale (EQ-VAS). The minimum score is 0 and maximum score is 100. (0) corresponds to " the worst health you can imagine", and the highest rate (100) corresponds to "the best health you can imagine".
Time Frame: Baseline, 6 weeks
Measure: Mean (Standard Deviation); unit: units
Arm/Group | IVIg Group | Placebo Group
Number analyzed (Participants) | 2 | 3
units | 15 (21.2) | 9.3 (22.8)

6. Secondary Outcome: Orthostatic Hypotension Symptom Assessment Questionnaire
Description: To determine the change in orthostatic Hypotension symptom (measured by the orthostatic hypotension symptom assessment questionnaire) measured at baseline and 6 weeks in individuals receiving IVIG. This is a 60 point orthostatic hypotenstion symptom assessment questionnaire. The minimum score possible is 0 and maximum is 60.
  Higher values represent worse outcome. We are reporting the total score.
Time Frame: Baseline, 6 weeks
Measure: Mean (Standard Deviation); unit: units
Arm/Group | Group A | Group B
Number analyzed (Participants) | 2 | 3
units | -9 (2.8) | 12 (9.5)

ADVERSE EVENTS:
Arm/Group | IVIg Group | Placebo Group
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/3
Other Adverse Events (participants affected / at risk) | 1/2 | 3/3
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IVIg Group (N=2) | Placebo Group (N=3)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1)
pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) — hand-foot skin reaction
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) — desquamation

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No